CLINICAL TRIAL: NCT01627171
Title: A Randomized Control Trial Comparing 4L PEGlyte to Regular Dose Pico-Salax and Split Dose Pico-Salax for Colonoscopy Bowel Preparation in Hospitalized Patients
Brief Title: Colonoscopy Preparation Optimization for INpatients- COIN Study
Acronym: COIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Khurram Khan, Assistant Professor of Medicine, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP 12-3657
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Endoscopy; Bowel Preparation Solutions
MeSH Terms: interventions — Bisacodyl; picosulfate sodium; Pico-Salax

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEG Lyte (Active Comparator): PEGlyte to be reconstituted with 4L of water and taken in the evening before the colonoscopy.
  Interventions: Drug: Bisacodyl 10mg; Drug: Polyethelene Glycol
- Pico Salax Split (Experimental): Two sachets of Pico-Salax with 1 taken the night before colonoscopy and the second taken the morning of colonoscopy.
  Interventions: Drug: Bisacodyl 10mg; Drug: Picosulfate sodium
- Pico Salax Night Before (Experimental): 2 sachets of Pico Salax mixed with water taken about 4 hours apart the night before colonoscopy
  Interventions: Drug: Bisacodyl 10mg; Drug: Picosulfate sodium

INTERVENTIONS:
Drug: Bisacodyl 10mg — Given at the start of the bowel preparation the day before colonoscopy
Drug: Polyethelene Glycol — 280g reconstituted in 4 liters of water
  Other Names: PEG-Lyte
  Arms: PEG Lyte
Drug: Picosulfate sodium — Two sachets, Each sachet has 10mg dose
  Other Names: Pico-Salax
  Arms: Pico Salax Night Before; Pico Salax Split

SUMMARY:
Colonoscopic examinations are performed routinely in hospitalized patients for a variety of indications. However, numerous limitations exist in hospitalized patients preventing an endoscopist from performing high quality examinations; possibly necessitating repeated procedures leading to increased cost and re-exposure to their inherent risks. One such prominent challenge lays in the adequacy of bowel cleansing. Inpatient status has been shown to be a predictor of poor bowel preparation as these patients are older, less mobile and have more co morbidities than the outpatient population. Currently, no standardized (or optimized) bowel preparation type or regimen for administration exists for the hospital inpatient population undergoing colonoscopy. Studies in the outpatient population have demonstrated that timing and choice of cathartic medication effects the cleanliness of the bowel preparation but there is no such clinical evidence for in-patients who receive whatever cathartic agent is on hospital formulary. The purpose of the study is compare efficacy, patient satisfaction, and adverse effects associated with low volume cathartic (Pico-Salax) to the current standard volume 4 liter (PEG-Lyte) and the effect of alternate timing of dosages.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient colonoscopy
* Age greater than 18 years old
* Able to give consent

Exclusion Criteria:

* No consent obtained
* Pregnancy or lactating
* Renal impairment
* Severe CHF (NYHA class 3/4)
* Recent myocardial infarction (preceding 6 months)
* Ileus
* Ascites
* Severe Colitis
* Toxic Megacolon
* Gastrointestinal Obstruction
* PEG tube
* Previous large bowel resection
* Allergy to study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Ottawa Bowel Prep Score | 30 minutes after procedure
  Using a standardized, validated score for measuring quality of bowel preparation

SECONDARY OUTCOMES:
Procedures Cancelled or repeated due to inadequate bowel preparation | During admission (average of 2 weeks)
  If bowel preparation is deemed inadequate to the point the procedure must be cancelled or rescheduled
Individual Components of Ottawa Bowel Prep Score | 30 minutes after procedure
  Each section of prep score evaluating the right, mid, and left colon, as well as the fluid score will be analyzed individually
Adverse Effects | Up to 48 hours after procedure
  Any adverse effects that may be attributed to the intervention
Tolerability of the preparation | Within 1 day of intervention
  A questionnaire to assess the overall tolerability of the preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Khurram J Khan, MD, BSc, Principal Investigator — St Josephs
Locations (1):
- St Joseph Hospital, Hamilton, Ontario, Canada